CLINICAL TRIAL: NCT04197128
Title: Comparative Evaluation of Novel Ribose Cross Linked Volumising Collagen Matrix v/s Ribose Cross Linked Resorbable Collagen Membrane and Bone Graft for Lateral Ridge Augmentation Around Implants: A Randomised Controlled Clinical Trial
Brief Title: Lateral Ridge Augmentation Around Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, Professor and Head of the Department, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02_D012_101329
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Alveolar Bone Resorption
Keywords: Lateral augmentation; Ribose cross-linked collagen; Dental Implant
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Intervention Model Description: The subjects are randomly divided into 2 groups i.e., Control and Test group each consisting of equal number of participants who are age and sex matched.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resorbable collagen membrane and bone graft (Active Comparator): Subjects will receive bovine derived bone graft and resorbable collagen membrane for augmentation.
  Interventions: Device: Resorbable Collagen membrane with bone graft for augmentation
- Ribose cross-linked collagen matrix (Experimental): Subjects will receive ribose cross linked collagen matrix for augmentation
  Interventions: Device: Ribose cross linked collagen matrix for augmentation

INTERVENTIONS:
Device: Resorbable Collagen membrane with bone graft for augmentation — Local anaesthesia Lignocaine and Adrenaline 1:80000 Injection (Lignox® 2% A, Indoco remedies Ltd, Mumbai) will be administered and midcrestal incison will be made and full thickness flap would be raised buccally. To obtain tension free adaptation of flap margins, the buccal flap advancement will be done using periosteal releasing incision. Implant osteotomies will be performed with sequential drilling and with standardised drills. All the subjects will receive the same implant system. (Norris medical ltd. Hatasia street, Nesher, Israel) For augmentation of deficient ridge, bovine bone graft will be place with overlying resorbable collagen membrane. Stabilisation would be achieved with internal resorbable horizontal mattress suture.
  The tension free flap margins will be adapted around the healing abutment with simple interrupted Vicryl 4.0, 3/8, reverse cutting resorbable sutures (Ethicon, Hamburg, Germany)
  Other Names: Cerabone®; Ossix Plus®
  Arms: Resorbable collagen membrane and bone graft
Device: Ribose cross linked collagen matrix for augmentation — Local anaesthesia Lignocaine and Adrenaline 1:80000 Injection (Lignox® 2% A, Indoco remedies Ltd, Mumbai) will be administered and midcrestal incison will be made and full thickness flap would be raised buccally. To obtain tension free adaptation of flap margins, the buccal flap advancement will be done using periosteal releasing incision.
  Implant osteotomies will be performed with sequential drilling and with standardised drills. All the subjects will receive the same implant system. (Norris medical ltd. Hatasia street, Nesher, Israel) For augmentation of deficient ridge, ribose cross linked collagen matrix will be cut and adapted to the buccal wall and ridge around the buccal aspect of healing abutment. Stabilisation would be achieved with internal resorbable horizontal mattress suture.
  The tension free flap margins will be adapted around the healing abutment with simple interrupted 4.0, 3/8, reverse cutting resorbable sutures (Ethicon, Hamburg, Germany).
  Other Names: Ossix Volumax®
  Arms: Ribose cross-linked collagen matrix

SUMMARY:
The rehabilitation of dentoalveolar defects and tooth loss has seen remarkable advancements over time. Extraction of tooth leads to reduction in physiologic dimension of bone and it is imperative to evaluate the site before implant placement. To overcome the loss of volume and to avoid complications, procedures to restore the resorbed alveolar bones prior to or during implant placement are usually performed.

Lateral bone augmentation procedures with guided bone regeneration (GBR) are well documented in the literature with predictable results. It generally involves bone substitute xenograft and bioresorbable membrane combined with implant placement in single stage procedure or separately in two- stage procedure. As the search for better and improved materials continues, a porcine derived ribose cross-linked volumising collagen matrix (VCMX) based on GLYMATRIX® technology has been introduced which showed benefits over the conventional membranes in terms of simplified procedure, degradation, membrane exposure and healing. The collagen scaffold has been reportedly used as a core material for guided bone regeneration, when there is sufficient bone to place an implant but a horizontal defect is present in the crestal ridge. As part of augmentation VCMX is designed to expand and ossify during healing. The advantage of the material is that when placed in one or two layers, it may eliminate the use of bone substitute or connective tissue graft thus simplifying the augmentation procedure. In addition, adding a bone substitute is a valid option based on indication.

In the quest of better material and simplified procedures, few authors have performed case studies based on application of VCMX for guided bone regeneration around dental implants and has shown promising results. However, there are no controlled clinical trials on application of VCMX for lateral ridge augmentation. Thus, the present study aims to assess the efficiency of VCMX compared to resorbable collagen membrane (RCM) and bone graft (BG) for lateral ridge augmentation around implants through a well designed, controlled clinical trial.

DETAILED DESCRIPTION:
Source of data Patient visiting the Outpatient Section of the Department of Periodontology, Krishnadevaraya College of Dental Sciences and Hospital for replacement of lost teeth will be screened and randomly recruited for the study as per inclusion and exclusion criteria. The eligible subjects will be informed of the nature and benefits of the participation of the study and a written signed consent will be obtained.

Method of collection of data Sample Size The study would be a prospective, randomized controlled clinical trial. A sample size of 28 subjects with equal number of males and females who are eligible as per the inclusion criteria, belonging to 20 - 50 years of age group would be considered for the study. Sample size is calculated using online software (OpenEpi) Open Source Epidemiologic Statistics for Public Health, Version 3.01. Estimation is done considering a similar previous study to acquire 80% power and 5% type 1 error in power calculation.

ELIGIBILITY:
Inclusion Criteria:

1. Cooperative patients willing to participate in the study belonging to 20-50 years of age group
2. Patients indicated for implant placement
3. Based on SAC classification (Straight forward, Advanced, Complex), if the bone defect has at least two walls intact and implant placement is possible within the confines of ridge.10 In the present study, subjects belonging to Advanced category i.e., where simultaneous guided bone regeneration and implant placement is possible it would be considered.
4. Full mouth plaque score (FMPS) < 20 %, Full mouth bleeding score (FMBS) < 20 %.11
5. Ability to comply with the study related procedures such as exercising good oral hygiene and attending all follow-up examinations.
6. Ability to fully understand the nature of the proposed surgery and ability to sign the informed consent form.

   -

Exclusion Criteria:

1. Smokers
2. Probing depth >4 mm
3. General contraindications for dental and/or surgical treatment
4. History of malignancy, radiotherapy, or chemotherapy for malignancy within the past 5 yrs
5. Pregnancy or breast feeding
6. Previous and concurrent medication affecting mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs)
7. History of any allergic diseases -

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-20 (Estimated)

PRIMARY OUTCOMES:
Ridge width | 6 months
  Ridge width would be measured pre-operatively and post-operatively using Cone beam computed tomography.
Gingival thickness | 6 months
  Clinical and radiographic assessment would be performed

SECONDARY OUTCOMES:
Patient- reported outcome 1 | 6 months
  Post operative pain and discomfort would be measured using Visual analogue scale
Patient reported outcome 2 | 6 months
  Number of analgesics consumed would be assessed during post- operative period
Safety evaluation 1 | 6 months
  Number of subjects with adverse healing
Safety evaluation 2 | 6 months
  Number of subjects who had membrane exposure

CONTACTS AND LOCATIONS:
Overall Officials: Prabhuji MLV, MDS, Study Director — Krishnadevaraya College of Dental Sciences; Karthikeyan Bangalore Varadhan, MDS, Study Director — Krishnadevaraya College of Dental Sciences
Locations (1):
- Krishnadevaraya College of Dental Sciences and Hospital, Bengaluru, Karnataka, India

REFERENCES:
- [Background] Friedmann A, Gissel K, Soudan M, Kleber BM, Pitaru S, Dietrich T. Randomized controlled trial on lateral augmentation using two collagen membranes: morphometric results on mineralized tissue compound. J Clin Periodontol. 2011 Jul;38(7):677-85. doi: 10.1111/j.1600-051X.2011.01738.x. Epub 2011 May 10. PMID 21557757
- [Background] Zubery Y, Nir E, Goldlust A. Ossification of a collagen membrane cross-linked by sugar: a human case series. J Periodontol. 2008 Jun;79(6):1101-7. doi: 10.1902/jop.2008.070421. PMID 18533790
- [Background] Smidt A, Gutmacher Z, Sharon E. A nouveau collagen scaffold to simplify lateral augmentation of deficient ridges between natural teeth. Quintessence Int. 2019;50(7):576-582. doi: 10.3290/j.qi.a42652. PMID 31161157